CLINICAL TRIAL: NCT01228032
Title: Improving Primary Care of Patients With Mental Disorders
Brief Title: The Health Outcomes Management and Evaluation (HOME) Study
Acronym: HOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Druss, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00027782; 2R01MH070437-06A1 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Hyperlipidemia; Heart Disease; High Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Heart Diseases; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Care team
- Control (No Intervention): referral only

INTERVENTIONS:
Other: Care team — The ICC will provide care for both the index cardiometabolic conditions and common acute and chronic comorbidities.
  Other Names: randomized control
  Arms: Intervention

SUMMARY:
There is an urgent need to develop practical, sustainable approaches to improving medical care for persons treated in community mental health settings. This study will test a novel approach for improving mental health consumers based on a partnership model between a Community Mental Health Center and a Community Health Center. When this study is completed, it will provide a model for a medical home for persons with severe mental illness that is clinically robust, and organizationally and financially sustainable

DETAILED DESCRIPTION:
Findings of excess cardiometabolic morbidity and mortality in persons with severe mental illness (SMI) have led to a growing interest by Community Mental Health Centers (CMHCs) in improving the medical care of the populations they treat. However, these organizations face a number of financial and organizational barriers to implementing and sustaining such programs. In previous and ongoing work, the study team has documented the promise of team-based models in improving health and health care in this population. This study will test a novel approach for improving mental health consumers based on a partnership model between a CMHC and a Community Health Center (CHC). This partnership will capitalize on collocation of services, the primary care expertise of the CHC, and favorable reimbursement conditions, to develop a program that is both clinically robust and financially and organizationally sustainable A total of 300 CMHC clients with a severe mental illness and one or more active cardiometabolic problem (diabetes, hypertension, hyperlipidemia) will be randomized to either onsite Integrated Community Care (ICC) (n=150) or to a referral to the partner community health center (CHC) (n=150) for their medical problems. For those in the ICC, the CHC will establish a satellite clinic at the CMHC staffed by a physician assistant and care manager. The ICC will provide care for both the index cardiometabolic conditions and common acute and chronic comorbidities.

The study will use standardized, validated instruments to assess the impact of integrated community care on quality and outcomes of cardiometabolic and general medical care. A budget impact analysis will be used to assess the program's financial and organizational sustainability. When this study is completed, it will provide a model for CMHCs to provide a medical home for the populations they serve.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Cobb County CSB
* one or more of the following conditions: hyperlipidemia, high blood pressure, heart failure, diabetes
* able to give consent

Exclusion Criteria:

* unable to give consent
* does not have a cardiometabolic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of healthcare services received | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Druss, MD MPH, Principal Investigator — Emory University
Locations (1):
- Cobb County Community Service Board, Marietta, Georgia, United States